CLINICAL TRIAL: NCT00628927
Title: An Evaluation of Neurocognitive Function, Oxidative Damage, and Their Association With Treatment Outcomes in Methamphetamine and Cocaine Abusers
Brief Title: An Eval of Neurocognitive Function, Oxidative Damage, and Their Association With Outcomes in METH and Cocaine Abusers.
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Theresa Winhusen, Associate Professor, University of Cincinnati
Other Study IDs: NIDA-CTN-0031A; 5U10DA013732 (NIH); U10DA013732 (NIH)
Record Dates: First submitted 2008-03-03; First posted 2008-03-05 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Stimulant Dependence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample for the oxidative stress/damage analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- METH and/or cocaine dependent group: The METH and/or cocaine dependent group were also enrolled in CTN0031 (NCT00573183) and seeking treatment. This group will be analyzed based on whether or not they completed treatment as defined by the study.
- Non METH and/or cocaine dependent group: The Non METH and/or cocaine dependent group participants are normal controls recruited from the community.

SUMMARY:
The purpose of this study is to determine whether performance on neurocognitive measures predicts treatment outcomes in individuals with substance abuse disorders. A second purpose is to compare the risk of damage, as well as actual damage, to DNA and other cell parts in people with substance abuse disorders to that of people who do not have substance abuse disorders.

DETAILED DESCRIPTION:
The primary objective of this study is to replicate the finding that performance on the Stroop color-word interference task is predictive of treatment completion in participants with cocaine use disorders and to extend this finding to participants with Methamphetamine use disorders. Secondary objectives include evaluating whether:

1. performance on various neurocognitive measures, including the Stroop, Rey Auditory-Verbal Learning Test (RAVLT), Iowa Gambling Task (GT), Wisconsin Card Sorting Task (WCST), the Barratt Impulsiveness Scale version -11 (BIS-11), and the Frontal Systems Behavior Scale (FrSBe) is predictive of treatment attrition and stimulant use outcomes in METH/cocaine abusers;
2. neurocognitive test performance is associated with oxidative damage, a severe consequence of oxidative stress, in METH/cocaine abusers;
3. oxidative damage is predictive of treatment attrition and substance use outcomes in METH/cocaine abusers,
4. oxidative damage in METH/cocaine abusers is significantly greater than that of a normal comparison group and
5. exploratory analyses reveal a significant relationship among oxidative stress, neurocognitive function, and treatment outcomes in METH/cocaine abusers.

ELIGIBILITY:
Inclusion Criteria (METH and/or Cocaine Dependent Group):

* be randomized into the CTN-0031 (STAGE-12) trial
* current abuse or dependence for METH and/or cocaine
* endorse METH and/or cocaine as the primary drug of choice
* able to correctly distinguish the colored stimuli on the Stoop task.

Exclusion Criteria (METH and/or Cocaine Dependent Group):

* history of stroke
* history of a seizure disorder

Inclusion Criteria (Non-METH and/or Cocaine Dependent Group):

* be 18 years of age or older
* be able to understand the study and provide written informed consent in English

Exclusion Criteria (Non-METH and/or Cocaine Dependent Group):

* history of stroke
* history of a seizure disorder
* positive urine toxicology screen
* screen positive for Major Depressive Syndrome, other Depressive Syndrome, Panic Syndrome, or other Anxiety Syndrome
* meet criteria for ADHD
* have HIV/AIDS
* history of an injury in which consciousness was lost for more than 30 minutes
* meet DSM-IV criteria for dependence (either current or lifetime) for any psychoactive substance other than nicotine or for abuse (both current and lifetime) for any psychoactive substance other than nicotine or for alcohol for which a life-time history of abuse is allowed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons randomized into the National Drug Abuse Treatment Clinical Trials Network STAGE-12 Study (CTN-0031- NCT00573183)
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Winhusen, Ph.D., Principal Investigator — University of Cincinnati
Locations (6):
- United States (6):
  - Gateway Community Services, Jacksonville, Florida
  - Maryhaven, Columbus, Ohio
  - Willamette Family Treatment Services, Eugene, Oregon
  - ChangePoint, Inc., Portland, Oregon
  - Nexus Recovery Center, Dallas, Texas
  - Recovery Centers of King County, Seattle, Washington

REFERENCES:
- [Result] Winhusen TM, Somoza EC, Lewis DF, Kropp FB, Horigian VE, Adinoff B. Frontal systems deficits in stimulant-dependent patients: evidence of pre-illness dysfunction and relationship to treatment response. Drug Alcohol Depend. 2013 Jan 1;127(1-3):94-100. doi: 10.1016/j.drugalcdep.2012.06.017. Epub 2012 Jul 6. PMID 22771145
- [Derived] Winhusen T, Walker J, Brigham G, Lewis D, Somoza E, Theobald J, Somoza V. Preliminary evaluation of a model of stimulant use, oxidative damage and executive dysfunction. Am J Drug Alcohol Abuse. 2013 Jul;39(4):227-34. doi: 10.3109/00952990.2013.798663. Epub 2013 Jun 28. PMID 23808868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As an ancillary study to CTN-0031, six of the nine sites participating in CTN-0031 were chosen to participate in the present study. At the participating sites, participants who were randomized into CTN-0031 were eligible to be screened for the present study. Normal controls were recruited via advertising from one study site.
Pre-assignment Details: 6 stimulant abusers met at least one exclusion criterion, 3 for a history of stroke and 3 for a history of seizures. 2 of those 6 were incorrectly enrolled into the study. The most common exclusion criteria met by the normal control screeners was having a DSM-IV substance use diagnosis and positive urine toxicology screen.
Groups:
- Simulant Dependent Participants: Stimulant Dependent pts entering treatment who are also enrolled in CTN0031
- Normal Control Participants: Normal Control participants recruited from the community
Period: Overall Study
Arm/Group | Simulant Dependent Participants | Normal Control Participants
Started | 183 | 30
Completed | 175 | 30
Not Completed | 8 | 0
Not completed — Problems performing blood draw | 6 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Equipment failure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Stimulant dependent participants were starting treatment, and participating in the CTN0031 study. Normal controls were recruited from the community.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simulant Dependent Participants | Normal Control Participants | Total
Number analyzed (Participants) | 183 | 30 | 213
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 183 | 30 | 213
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (9.3) | 44.5 (9.5) | 39.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 17 | 142
  Male | 58 | 13 | 71
Region of Enrollment [Number; unit: participants]
  United States | 183 | 30 | 213

OUTCOME MEASURES:

1. Primary Outcome: Stroop Color-word Task
Description: The primary objective of this study was to replicate the finding that performance on the Stroop color-word interference task is predictive of treatment completion in participants with cocaine use disorders (Streeter et al., 2007) and to extend this finding to participants with methamphetamine use disorders. In the Stroop, the participant is required to name the color of the ink in which a word is printed while inhibiting the overlearned response of reading the word (e.g., the word ''red'' might be printed in blue ink). The number of errors were subtracted from the time required (RT; Reaction Time) for each of the 3 trials, yielding three summary scores. The derived interference score is obtained by subtracting the RT for the first trial from the RT for the third trial.
Time Frame: Single study visit
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Stimulant Dependent Completers: Completers were those who attended the first 5 weeks of treatment without missing two or more consecutive weeks; a participant who attended the first 4 weeks of treatment and missed the fifth week was considered a treatment completer if s/he attended treatment during the sixth week
- Stimulant Dependent Treatment Non-Completers: Non-completers were those who failed to attend the first 5 weeks of treatment without missing two or more consecutive weeks; alternately, a participant who attended the first 4 weeks of treatment and missed the fifth week was considered a treatment non-completer if s/he did not attend treatment during the sixth week Data for the two ineligible but enrolled participants was removed from the analysis.
Arm/Group | Stimulant Dependent Completers | Stimulant Dependent Treatment Non-Completers
Number analyzed (Participants) | 130 | 51
seconds | 55.4 (22.9) | 50.5 (21.0)

2. Secondary Outcome: Barrett Impulsiveness Scale Version 11 (BIS-11)
Description: The BIS-11 consists of 30 self-report items, with responses in a four-point Likert-type scale (0 - 3)ranging from "Rarely/Never" to "Almost Always/Always" and comprises three domains: Attentional impulsiveness (AI), Motor impulsiveness (MI), and Non-planning impulsiveness (NP); these three domains are summed to yield a total score; higher scores reflect greater impulsivity. The total score was utilized as the BIS-11 predictor measure (possible score range 0 - 90).
Time Frame: Single study visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Stimulant Dependent Completers: Completers were those who attended the first 5 weeks of treatment without missing two or more consecutive weeks; a participant who attended the first 4 weeks of treatment and missed the fifth week was considered a treatment completer if s/he attended treatment during the sixth week Data from one participant was excluded from analysis due to lack of completeness
- Stimulant Dependent Treatment Non-Completers: Non-completers were those who failed to attend the first 5 weeks of treatment without missing two or more consecutive weeks; alternately, a participant who attended the first 4 weeks of treatment and missed the fifth week was considered a treatment non-completer if s/he did not attend treatment during the sixth week Data from the two ineligible by enrolled participants was removed from the analysis.
  Data from 3 other participants was incomplete and therefore removed from the analysis.
Arm/Group | Stimulant Dependent Completers | Stimulant Dependent Treatment Non-Completers
Number analyzed (Participants) | 129 | 48
units on a scale | 66.7 (9.3) | 69.4 (7.5)

3. Secondary Outcome: Tail Length From the Comet Assay for Oxidative Damage
Description: The test for oxidative damage was derived from a blood sample which was analyzed for tail length from the comet assay; higher scores reflect greater oxidative damage.
Time Frame: Single study visit
Measure: Mean (Standard Deviation); unit: µm
Groups:
- Stimulant Dependent Completers: Completers were those who attended the first 5 weeks of treatment without missing two or more consecutive weeks; a participant who attended the first 4 weeks of treatment and missed the fifth week was considered a treatment completer if s/he attended treatment during the sixth week 3 participant samples were insufficient for analysis
- Stimulant Dependent Treatment Non-Completers: Non-completers were those who failed to attend the first 5 weeks of treatment without missing two or more consecutive weeks; alternately, a participant who attended the first 4 weeks of treatment and missed the fifth week was considered a treatment non-completer if s/he did not attend treatment during the sixth week Data for 2 participants who were ineligible but enrolled were removed from analysis 1 participant did not complete the blood draw
  1 participant sample was insufficient for analysis
- Normal Controls: Normal controls recruited from the community.
Arm/Group | Stimulant Dependent Completers | Stimulant Dependent Treatment Non-Completers | Normal Controls
Number analyzed (Participants) | 127 | 49 | 30
µm | 17.3 (10.1) | 15.6 (8.5) | 16.5 (7.2)

ADVERSE EVENTS:
Arm/Group | Simulant Dependent Participants | Normal Control Participants
Serious Adverse Events (participants affected / at risk) | 0/175 | 0/30
Other Adverse Events (participants affected / at risk) | 0/175 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No